CLINICAL TRIAL: NCT05636917
Title: Study of the Diagnostic Accuracy of the Slump and Straight Leg Raise Neurodynamic Tests in Patients With Clinical Suspicion of Lumbar Radiculopathy
Brief Title: Study of the Diagnostic Accuracy of the Neurodynamic Tests in Patients With Lumbar Radiculopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Alberto Montaner Cuello, Principal Investigator, Universidad de Zaragoza
Other Study IDs: PI21/073
Record Dates: First submitted 2022-10-25; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Lumbar Radiculopathy
Keywords: Nerve Root Disorder; Neurodynamics Test; Diagnostic Accuracy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- radiculopathy: Patients with suspected radiculopathy who are prescribed the nerve conduction test at the Lozano-Blesa University Hospital and who have undergone or are awaiting an MRI scan.

SUMMARY:
Lumbar radiculopathy is a relevant cause of disability and morbidity, accounting for between 23 and 57% of the cases of patients with low back pain and representing a significant expense due to the sick leave and health care that may be required.

Nuclear magnetic resonance and electromyography are the most commonly used tests for the diagnosis of the pathology.

Neurodynamic tests represent a sequence of structured movements with the purpose of increasing the mechanical stress of the neural tissue. These tests are currently an important aspect of the physical examination of the patient when there is suspicion of neural involvement, allowing the physiological and mechanical capacities of the nerve to be evaluated.

The Slump and Straight Leg Raise neurodynamic tests are the two best known tests for assessing the mechanosensitivity of the sciatic nerve and its component roots.

The hypothesis of this observational study is that the straight leg raising and Slump neurodynamic tests with precise diagnostic criteria are valid tools for the diagnosis of lumbar radiculopathy.

DETAILED DESCRIPTION:
Background and justification Background Lumbar radiculopathy is a relevant cause of disability and morbidity and may constitute between 23 and 57% of the cases of patients with low back pain and represents an important expense due to the sick leave and health care that may be required. It is a pathological process that can affect different lumbar roots and can cause radiating symptoms that manifest in the territory of the lower limb that includes this root. Some studies estimate the prevalence in the general population to be between 1.6 and 13.4%, with the predominant age range being between 45 and 64 years of age and affecting men more frequently than women.

Protrusion or migration of the lumbar intervertebral disc is the most common cause of nerve root irritation and subsequent radiculopathy. Disc herniation is define as a localised displacement of disc material beyond the normal margins of the intervertebral disc space resulting in pain, weakness or numbness in a myotomal or dermatomal distribution.

In clinical practice, the diagnosis of lumbar radiculopathy involves the use of several tools and procedures including neuropathic pain screening, clinical neurological examination, electro-diagnostic, nerve root block and radiological imaging. The gold standard for the diagnosis of lumbar disc herniation is surgery; however, when assessing the validity of subjective tests or physical examination findings, the use of cross-sectional imaging as a gold standard may be considered an acceptable substitute, always bearing in mind that the results of any imaging test should be closely correlated with the clinical examination.

Many clinical guidelines advise muscle strength testing, sensory testing and different neurodynamic tests for the diagnosis of lumbar disc herniation with radiculopathy.

Neurodynamic tests represent a structured sequence of movements aimed at increasing the mechanical stress on the neural tissue, and are now an important aspect of the physical examination of the patient when there is suspicion of neural involvement, allowing assessment of the physiological and mechanical capabilities of the nerve. These neurodynamic tests include the mechanism of structural differentiation that allows a specific assessment of neural tissue and makes it possible to rule out a musculoskeletal origin of the patient's symptoms.

When used in isolation, the diagnostic performance of most physical tests (muscle weakness or paresis, muscle atrophy, impaired reflexes, sensory deficits) is poor. Some tests (forward flexion, hyperextension test and Slump test) perform slightly better, but the number of studies is small.

Rapid and accurate clinical diagnosis is essential in the management of these patients in order to decide on the correct treatment.

Justification The clinical manifestations caused by a herniated disc are derived from the possible involvement of the nerve root, and neurodynamic tests could presumably help us to detect the pathology by testing neural mechano-sensitivity. Neurodynamic tests are interpreted using structural differentiation, range of motion and sensory responses as the location or quality of symptoms in relation to the contralateral limb and compared with normalisation results in healthy populations. However, existing studies of the Straight Leg Raise test are not very sensitive and those of the Slump test with better sensitivity results are very scarce.

Once symptoms compatible with nerve root involvement due to disc herniation are found, the test of choice to diagnose the pathology is magnetic resonance imaging. Nerve conduction tests are also effective to see the real neural involvement that radiculopathy may be causing, but these complementary tests may take a long time or even be inaccessible, and early treatment may be essential.

The two neurodynamic tests that have been shown to modify tension and/or generate forces on lumbar nerve roots are the Straight Leg Raise test and the Slump test. However, many studies to date have concluded that these tests have low sensitivity and specificity. The causes of this low validity could be the ambiguity of the diagnostic criteria including the modification of symptoms with structural differentiation, which is essential for a correct interpretation of the test and subsequent diagnostic suspicion. Most existing studies on the diagnostic accuracy of these neurodynamic tests do not include structural differentiation in their diagnostic criteria.

However, neurodynamic tests are an affordable, simple and quick tool available to all clinicians trained in neurodynamics. By defining the diagnostic criteria more precisely and using magnetic resonance imaging as the gold standard, the validity of these neurodynamic tests could be improved, making them useful diagnostic tools in clinical contexts.

A rapid diagnosis could ensure the good evolution of the patient by reducing the time to decide on the treatment to be carried out.

Hypothesis The Neurodynamic Straight Leg Raise and Slump tests with precise diagnostic criteria are valid tools for the diagnosis of lumbar radiculopathy.

Objectives Main objective To study the diagnostic accuracy of the Slump and Straight Leg Raise neurodynamic tests in patients with lumbar radiculopathy.

Secondary objectives

* To analyse the diagnostic accuracy of the Slump test with structural differentiation in the detection of lumbar radiculopathy.
* To analyse the diagnostic accuracy of the straight leg raise test in the detection of lumbar radiculopathy.
* To compare the diagnostic accuracy of the Slump test versus the Straight Leg Raise test in this pathology.
* To study the diagnostic validity of the Slump test including nerve conduction tests together with the standard MRI pattern.

Procedure The patient who is prescribed the nerve conduction test and who has undergone or is awaiting an MRI scan will be informed of the possibility of participating in the study and those who agree to participate voluntarily will sign the informed consent form.

Once the consent has been signed, data will be collected from the patient's clinical history. The assessor will take the data from the patient's history and exclude those who do not meet the inclusion/exclusion criteria. Age, sex, weight and height shall be recorded in the medical record.

The assessor will perform the neurodynamic straight leg raise test with the Bragard manoeuvre, the Slump test and the modified Slump test. In addition, each patient will complete the pain scales for neuropathic pain assessment (DN4), the Oswestry Low Back Pain Disability Scale and the Visual Analogue Scale (VAS), recording the data from these tests.

The physiotherapist in charge of performing the tests will not know the results of the imaging tests.

The Straight Leg Raise test or also known as the Lasègue test is performed with the patient in the supine position and, without moving the spine, the leg is passively raised while maintaining knee extension until symptoms appear. The test is considered positive if the patient does not reach an amplitude of 70° of hip flexion and this amplitude is different with respect to the other limb, no structural differentiation is specified to rule out muscular structures. The classic Lasegue test repeated the manoeuvre with knee flexion and hip flexion, and was considered positive if the second manoeuvre did not reproduce the symptoms and the first did. In the study the investigators will perform the Straight Leg Raise test with the addition of the Bragard manoeuvre which involves dorsiflexion of the ankle and involves more pretension of the neural system and with structural differentiation.

The Slump test adds tension on all lumbar nerve roots and includes the mechanism of structural differentiation as opposed to the classic Straight Leg Raise test. The test is performed in a seated position, with flexion of the cervical, dorsal and lumbar spine. The physiotherapist extends the patient's knee to the presence of symptoms and, depending on the region of symptoms, a remote joint movement is performed to establish a differential diagnosis between pain of musculoskeletal origin and pain of neural origin. The modified Slump test to further pretension the sciatic nerve involves maximum lumbar flexion, contralateral lumbar tilt of the roots to be assessed and internal hip rotation of the homolateral limb.

Diagnostic criteria for neurodynamic tests. The test is considered positive if the structural differentiation is positive and any of these criteria are met:

* It reproduces the patient's symptoms.
* It produces symptoms with decreased range of motion with respect to the other limb.
* It produces symptoms with asymmetry in the location or type of symptom perceived with respect to the other limb.

Statistical analysis All data analysis will be performed with IBM SPSS Statistics (Version 21.0.0.0). For the descriptive analysis of quantitative variables, indices of central tendency and indices of dispersion will be used. For qualitative variables, a study of frequencies will be carried out to find out what percentage of them are present.

Prior to the study, quantitative variables will be analysed to determine normality using the Kolmogorov-Smirnov test.

For the validity study, the sensitivity, specificity, predictive values and probability ratios of the Slump test and the Straight Leg Raise test will be calculated. Contingency tables 2x2 will be drawn up for the results of each of the tests, with their diagnostic criteria, with the MRI and electrophysiological tests. A 95% confidence interval will be established for these values.

Ethical aspects The study to be carried out does not involve any invasive procedure and does not pose any risk to the subjects participating in it. In the performance of the neurodynamic tests, the symptoms that the patient already has due to the neural response of the test can be reproduced.

Subject data will be coded in such a way that no personal patient data will be included in the study database and no one other than the investigators will have access to the database.

Participants will not receive financial or other compensation for their participation in the study.

All participants will be informed in writing, by means of an information sheet, and will be required to sign the informed consent form.

Timeline The project will start once it receives the approval of the Clinical Research Ethics Committee of Aragon (Spain). Subjects will be scheduled according to their availability and that of the investigators. Fieldwork is expected to last 1-2 years. Subsequently, data will be analysed and published in an estimated period of 1 year.

Budget The project has no funding. The materials used belong to the principal investigator and the clinical neurophysiology service of the Hospital Clínico Universitario Lozano Blesa located in the city of Zaragoza (Aragón, Spain).

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 75 years of age.
* Having symptoms compatible with lumbar radiculopathy at the time of the study. Intermittent or constant pain in the lumbar area or radiating to a distal extremity, to the gluteal fold; or distribution of pain in all or part of the dermatomic area of one or two adjacent lumbosacral nerve roots (L3-S2 segments).
* Have undergone or are awaiting MRI of the lumbar region.
* Have been referred for an electrophysiological study of the sciatic nerve or its branches.
* Have sufficient comprehension and communication skills to be able to communicate their symptoms and their characteristics.
* Accept and give their consent to participate voluntarily in the study and provide their clinical data anonymously.

Exclusion Criteria:

* Having radiological tests with a diagnosis of spondylolysis and/or spondylolisthesis in the lumbar region.
* Having been diagnosed with diabetes, thyroid dysfunction, rheumatoid arthritis, heart and/or lung disease, alcoholism, HIV+, herpes zoster infection, multiple sclerosis, hereditary neuropathy or any known neurodegenerative disease and/or pregnancy.
* Have undergone lumbar surgery and/or transforaminal epidural steroid injection within the previous 12 months.
* Have received physiotherapeutic neurodynamic treatment.
* Have suffered a fracture of any vertebrae of the spine.
* Have been diagnosed with other compressive causes or causes that produce irritation of the lumbar roots or stenosis of the spinal canal.
* Be unable or have contraindications to adopt the supine decubitus and/or seated position with lumbar, dorsal and cervical flexion or to maintain the position for the duration of the tests.
* Present any physical contraindication (red flags) such as neoplastic processes, serious infections; or psychological contraindication (yellow flags) such as psychiatric pathologies that could influence the state of the subjects or the results of the study.
* That the MRI is performed more than 12 months after the clinical examination.
* Failure to complete all the assessment phases of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample is recruited from among individuals pending nerve conduction testing for suspected lumbar radiculopathy and who have undergone or are pending lumbar MRI. Subjects will be included in the sample using the consecutive case sampling method which avoids overestimation of the diagnostic accuracy of the test to be studied.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09-04 (Estimated)

PRIMARY OUTCOMES:
Disc injuries | Through study completion, an average of 1 year
  Quantify by nuclear magnetic resonance whether and to what extent the disc is damaged.
Nerve conduction tests. Electromyography. | Through study completion, an average of 1 year
  Electromyography are performed to assess nerve root status. The electromyography result shall be classified according to the specialist's report. The items are "Mild radiculopathy" and "Severe radiculopathy"
Straight leg raise test | Through study completion, an average of 1 year
  Straight leg raise test is performed to assess the mechanosensitivity of the nerve.
Slump test | Through study completion, an average of 1 year
  Slump test is performed to assess the mechanosensitivity of the nerve.
Pain scales | Through study completion, an average of 1 year
  The Visual Analogue Scale is used to assess the patient's level of impairment (VAS). Values from 0 to 10. 0 no pain, 10 maximum pain.
DN4 Neuropathic pain questionnaire. | Through study completion, an average of 1 year
  The DN4 questionnaire consists of a total of 10 items grouped in 4 sections. The first seven items are related to the quality of pain (burning, painful, cold, electric shocks) and its association to abnormal sensations (tingling, pins and needles, numbness, itching).The other 3 items are related to neurological examination in the painful area (touch hypoesthesia, pinprick hypoesthesia, tactile allodynia). A score of 1 is given to each positive item and a score of 0 to each negative item. The total score is calculated as the sum of all 10 items, and the cut-off value for the diagnosis of neuropathic pain is a total score of 4/10.
The Oswestry scale | Through study completion, an average of 1 year
  The Oswestry scale is used to assess the patient's level of impairment. Shows the percentage of dysfunction. The total score is expressed as a percentage (from 0 to 100 %). Higher values describe greater functional limitation. Between 0-20 %: minimal functional limitation; 20-40 %: moderate; 40-60 %: severe; 60-80 %: disability; and above 80 %: maximum functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Bueno-Gracia, PT PhD, Study Director — Universidad Zaragoza; Santos Caudevilla-Polo, PT PhD, Study Director — Universidad Zaragoza
Locations (1):
- Alberto Montaner Cuello, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruschel LG, Agnoletto GJ, Aragao A, Duarte JS, de Oliveira MF, Teles AR. Lumbar disc herniation with contralateral radiculopathy: a systematic review on pathophysiology and surgical strategies. Neurosurg Rev. 2021 Apr;44(2):1071-1081. doi: 10.1007/s10143-020-01294-3. Epub 2020 Apr 13. PMID 32281018
- [Background] Tawa N, Rhoda A, Diener I. Accuracy of clinical neurological examination in diagnosing lumbo-sacral radiculopathy: a systematic literature review. BMC Musculoskelet Disord. 2017 Feb 23;18(1):93. doi: 10.1186/s12891-016-1383-2. PMID 28231784
- [Background] Beynon R, Elwenspoek MMC, Sheppard A, Higgins JN, Kolias AG, Laing RJ, Whiting P, Hollingworth W. The utility of diagnostic selective nerve root blocks in the management of patients with lumbar radiculopathy: a systematic review. BMJ Open. 2019 Apr 20;9(4):e025790. doi: 10.1136/bmjopen-2018-025790. PMID 31005925
- [Background] Clark R, Weber RP, Kahwati L. Surgical Management of Lumbar Radiculopathy: a Systematic Review. J Gen Intern Med. 2020 Mar;35(3):855-864. doi: 10.1007/s11606-019-05476-8. Epub 2019 Nov 11. PMID 31713029
- [Background] Scaia V, Baxter D, Cook C. The pain provocation-based straight leg raise test for diagnosis of lumbar disc herniation, lumbar radiculopathy, and/or sciatica: a systematic review of clinical utility. J Back Musculoskelet Rehabil. 2012;25(4):215-23. doi: 10.3233/BMR-2012-0339. PMID 23220802
- [Background] Kreiner DS, Hwang SW, Easa JE, Resnick DK, Baisden JL, Bess S, Cho CH, DePalma MJ, Dougherty P 2nd, Fernand R, Ghiselli G, Hanna AS, Lamer T, Lisi AJ, Mazanec DJ, Meagher RJ, Nucci RC, Patel RD, Sembrano JN, Sharma AK, Summers JT, Taleghani CK, Tontz WL Jr, Toton JF; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of lumbar disc herniation with radiculopathy. Spine J. 2014 Jan;14(1):180-91. doi: 10.1016/j.spinee.2013.08.003. Epub 2013 Nov 14. PMID 24239490
- [Background] Joshi KC, Eapen C, Kumar SP. Normal sensory and range of motion (ROM) responses during Thoracic Slump Test (ST) in asymptomatic subjects. J Man Manip Ther. 2013 Feb;21(1):24-32. doi: 10.1179/2042618612Y.0000000015. PMID 24421610
- [Background] Shacklock M. Improving application of neurodynamic (neural tension) testing and treatments: a message to researchers and clinicians. Man Ther. 2005 Aug;10(3):175-9. doi: 10.1016/j.math.2005.03.001. Epub 2005 Apr 20. No abstract available. PMID 16038853
- [Background] Coppieters MW, Alshami AM, Babri AS, Souvlis T, Kippers V, Hodges PW. Strain and excursion of the sciatic, tibial, and plantar nerves during a modified straight leg raising test. J Orthop Res. 2006 Sep;24(9):1883-9. doi: 10.1002/jor.20210. PMID 16838375
- [Background] Coppieters MW, Butler DS. Do 'sliders' slide and 'tensioners' tension? An analysis of neurodynamic techniques and considerations regarding their application. Man Ther. 2008 Jun;13(3):213-21. doi: 10.1016/j.math.2006.12.008. Epub 2007 Mar 30. PMID 17398140
- [Background] Pesonen J, Shacklock M, Suomalainen JS, Karttunen L, Maki J, Airaksinen O, Rade M. Extending the straight leg raise test for improved clinical evaluation of sciatica: validity and diagnostic performance with reference to the magnetic resonance imaging. BMC Musculoskelet Disord. 2021 Sep 21;22(1):808. doi: 10.1186/s12891-021-04649-z. PMID 34548049
- [Background] Butler DS. Adverse mechanical tension in the nervous system: a model for assessment and treatment. Aust J Physiother. 1989;35(4):227-38. doi: 10.1016/S0004-9514(14)60511-0. PMID 25025621
- [Background] van der Windt DA, Simons E, Riphagen II, Ammendolia C, Verhagen AP, Laslett M, Deville W, Deyo RA, Bouter LM, de Vet HC, Aertgeerts B. Physical examination for lumbar radiculopathy due to disc herniation in patients with low-back pain. Cochrane Database Syst Rev. 2010 Feb 17;(2):CD007431. doi: 10.1002/14651858.CD007431.pub2. PMID 20166095
- [Background] Elvey RL. Physical evaluation of the peripheral nervous system in disorders of pain and dysfunction. J Hand Ther. 1997 Apr-Jun;10(2):122-9. doi: 10.1016/s0894-1130(97)80066-x. PMID 9188031
- [Background] Boyd BS, Villa PS. Normal inter-limb differences during the straight leg raise neurodynamic test: a cross sectional study. BMC Musculoskelet Disord. 2012 Dec 10;13:245. doi: 10.1186/1471-2474-13-245. PMID 23227972
- [Background] Lohkamp M, Small K. Normal response to Upper Limb Neurodynamic Test 1 and 2A. Man Ther. 2011 Apr;16(2):125-30. doi: 10.1016/j.math.2010.07.008. Epub 2010 Sep 1. No abstract available. PMID 20810302
- [Background] Nee RJ, Jull GA, Vicenzino B, Coppieters MW. The validity of upper-limb neurodynamic tests for detecting peripheral neuropathic pain. J Orthop Sports Phys Ther. 2012 May;42(5):413-24. doi: 10.2519/jospt.2012.3988. Epub 2012 Mar 8. PMID 22402638
- [Background] Majlesi J, Togay H, Unalan H, Toprak S. The sensitivity and specificity of the Slump and the Straight Leg Raising tests in patients with lumbar disc herniation. J Clin Rheumatol. 2008 Apr;14(2):87-91. doi: 10.1097/RHU.0b013e31816b2f99. PMID 18391677
- [Background] Ekedahl H, Jonsson B, Annertz M, Frobell RB. Accuracy of Clinical Tests in Detecting Disk Herniation and Nerve Root Compression in Subjects With Lumbar Radicular Symptoms. Arch Phys Med Rehabil. 2018 Apr;99(4):726-735. doi: 10.1016/j.apmr.2017.11.006. Epub 2017 Dec 15. PMID 29253501
- [Background] Yousif S, Musa A, Ahmed A, Abdelhai A. Correlation between Findings in Physical Examination, Magnetic Resonance Imaging, and Nerve Conduction Studies in Lumbosacral Radiculopathy Caused by Lumbar Intervertebral Disc Herniation. Adv Orthop. 2020 Jan 24;2020:9719813. doi: 10.1155/2020/9719813. eCollection 2020. PMID 32082626
- [Background] Gilbert KK, Brismee JM, Collins DL, James CR, Shah RV, Sawyer SF, Sizer PS Jr. 2006 Young Investigator Award Winner: lumbosacral nerve root displacement and strain: part 2. A comparison of 2 straight leg raise conditions in unembalmed cadavers. Spine (Phila Pa 1976). 2007 Jun 15;32(14):1521-5. doi: 10.1097/BRS.0b013e318067dd72. PMID 17572622
- [Background] Gilbert KK, Brismee JM, Collins DL, James CR, Shah RV, Sawyer SF, Sizer PS Jr. 2006 Young Investigator Award Winner: lumbosacral nerve root displacement and strain: part 1. A novel measurement technique during straight leg raise in unembalmed cadavers. Spine (Phila Pa 1976). 2007 Jun 15;32(14):1513-20. doi: 10.1097/BRS.0b013e318067dd55. PMID 17572621
- [Background] Coppieters MW, Crooke JL, Lawrenson PR, Khoo SJ, Skulstad T, Bet-Or Y. A modified straight leg raise test to differentiate between sural nerve pathology and Achilles tendinopathy. A cross-sectional cadaver study. Man Ther. 2015 Aug;20(4):587-91. doi: 10.1016/j.math.2015.01.013. Epub 2015 Jan 31. PMID 25680573
- [Background] Lai WH, Shih YF, Lin PL, Chen WY, Ma HL. Normal neurodynamic responses of the femoral slump test. Man Ther. 2012 Apr;17(2):126-32. doi: 10.1016/j.math.2011.10.003. Epub 2011 Nov 6. PMID 22056894
- [Background] Whiting PF, Rutjes AW, Westwood ME, Mallett S, Deeks JJ, Reitsma JB, Leeflang MM, Sterne JA, Bossuyt PM; QUADAS-2 Group. QUADAS-2: a revised tool for the quality assessment of diagnostic accuracy studies. Ann Intern Med. 2011 Oct 18;155(8):529-36. doi: 10.7326/0003-4819-155-8-201110180-00009. PMID 22007046
- [Background] Trainor K, Pinnington MA. Reliability and diagnostic validity of the slump knee bend neurodynamic test for upper/mid lumbar nerve root compression: a pilot study. Physiotherapy. 2011 Mar;97(1):59-64. doi: 10.1016/j.physio.2010.05.004. Epub 2010 Aug 1. PMID 21295239
- [Background] Gonzalez Espinosa de Los Monteros FJ, Gonzalez-Medina G, Ardila EMG, Mansilla JR, Exposito JP, Ruiz PO. Use of Neurodynamic or Orthopedic Tension Tests for the Diagnosis of Lumbar and Lumbosacral Radiculopathies: Study of the Diagnostic Validity. Int J Environ Res Public Health. 2020 Sep 26;17(19):7046. doi: 10.3390/ijerph17197046. PMID 32993094
- [Background] Bueno-Gracia E, Tricas-Moreno JM, Fanlo-Mazas P, Malo-Urries M, Haddad-Garay M, Estebanez-de-Miguel E, Hidalgo-Garcia C, Krauss JR. Validity of the Upper Limb Neurodynamic Test 1 for the diagnosis of Carpal Tunnel Syndrome. The role of structural differentiation. Man Ther. 2016 Apr;22:190-5. doi: 10.1016/j.math.2015.12.007. Epub 2015 Dec 23. PMID 26783037
- [Background] Urban LM, MacNeil BJ. Diagnostic Accuracy of the Slump Test for Identifying Neuropathic Pain in the Lower Limb. J Orthop Sports Phys Ther. 2015 Aug;45(8):596-603. doi: 10.2519/jospt.2015.5414. Epub 2015 Jun 24. PMID 26107044
- [Background] Perez C, Galvez R, Huelbes S, Insausti J, Bouhassira D, Diaz S, Rejas J. Validity and reliability of the Spanish version of the DN4 (Douleur Neuropathique 4 questions) questionnaire for differential diagnosis of pain syndromes associated to a neuropathic or somatic component. Health Qual Life Outcomes. 2007 Dec 4;5:66. doi: 10.1186/1477-7525-5-66. PMID 18053212
- [Background] Pomares Avalos AJ, Lopez Fernandez R, Zaldivar Perez DF. [Validation of the Oswestry disability scale for low back pain in patients with chronic back pain. Cienfuegos, 2017-2018]. Rehabilitacion (Madr). 2020 Jan-Mar;54(1):25-30. doi: 10.1016/j.rh.2019.10.003. Epub 2019 Dec 24. Spanish. PMID 32007179
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Shacklock M, Yee B, Van Hoof T, Foley R, Boddie K, Lacey E, Poley JB, Rade M, Kankaanpaa M, Kroger H, Airaksinen O. Slump Test: Effect of Contralateral Knee Extension on Response Sensations in Asymptomatic Subjects and Cadaver Study. Spine (Phila Pa 1976). 2016 Feb;41(4):E205-10. doi: 10.1097/BRS.0000000000001218. PMID 26571159
- [Background] Herrington L, Bendix K, Cornwell C, Fielden N, Hankey K. What is the normal response to structural differentiation within the slump and straight leg raise tests? Man Ther. 2008 Aug;13(4):289-94. doi: 10.1016/j.math.2007.01.013. Epub 2007 Mar 29. PMID 17395520
- [Background] Jaeschke R, Guyatt GH, Sackett DL. Users' guides to the medical literature. III. How to use an article about a diagnostic test. B. What are the results and will they help me in caring for my patients? The Evidence-Based Medicine Working Group. JAMA. 1994 Mar 2;271(9):703-7. doi: 10.1001/jama.271.9.703. No abstract available. PMID 8309035
- [Background] Shacklock M. Neurodynamics. Physiotherapy. 1995;81(1):9-16.
- [Background] Butler DS. The sensitive nervous system. 1st ed. Adelaide, Australia: NoigroupPublications; 2000
- [Background] Seoane T, Martín JLR, Martín-Sánchez E, Lurueña-Segovia S, Alonso Moreno FJ.Capítulo 5: Selección de la muestra: técnicas de muestreo y tamaño muestral.Semergen [Internet]. 2007;33(7):358-61. Available from: http://dx.doi.org/10.1016/S1138-3593(07)73915-1
- [Background] Cleland J. Netter. Exploración clínica en ortopedia. Un enfoque para fisioterapeutasbasado en la evidencia. 13th ed. Barcelona: Masson, S.A.; 2006. 528 p.